CLINICAL TRIAL: NCT02245672
Title: A Randomized, Double-blind, Double Dummy, Parallel Group Study to Determine the Local Equivalence of Multiple Doses of MGR001 to Advair Diskus Administered Via Oral Inhalation in Adult Asthma Patients
Brief Title: MGR001 / Advair Diskus Local Equivalence Study in Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mylan Pharma UK Ltd. (Industry)
Responsible Party: Sponsor
Organization: Viatris Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MGR001-3001
Record Dates: First submitted 2014-09-15; First posted 2014-09-19 (Estimated); Results first posted 2021-01-12 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: Asthma
Keywords: Asthma; fluticasone; salmeterol; CRC749; Diskus; Advair; FEV1; MGR001
MeSH Terms: conditions — Asthma | interventions — Salmeterol Xinafoate; Fluticasone-Salmeterol Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- MGR001 (Experimental): MGR001 administered two times per day by inhalation throughout the study
  Interventions: Drug: MGR001 (Fixed dose combination of Fluticasone propionate and salmeterol xinafoate)
- Advair Diskus (Active Comparator): Advair Diskus administered two times per day by inhalation throughout the study
  Interventions: Drug: Advair (Fixed dose combination of Fluticasone propionate and salmeterol xinafoate)
- Placebo (Placebo Comparator): Placebo for Advair Diskus and MGR001 administered two times per day by inhalation throughout the study
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MGR001 (Fixed dose combination of Fluticasone propionate and salmeterol xinafoate) — Fluticasone propionate (100 mcg) and salmeterol xinafoate (50 mcg) administered via the CRC749 inhaler device
  Arms: MGR001
Drug: Advair (Fixed dose combination of Fluticasone propionate and salmeterol xinafoate) — Fluticasone propionate (100 mcg) and salmeterol xinafoate (50 mcg) administered via the Diskus inhaler device
  Arms: Advair Diskus
Drug: Placebo — Placebo administered via the CRC749 and Diskus devices
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether MGR001 is equivalent to Advair Diskus when administered by inhalation in adult asthma patients

ELIGIBILITY:
Key inclusion criteria include:

* Male or female subjects aged ≥18 years. Females may be of either childbearing or non-childbearing potential
* Physician diagnosed history of asthma for at least 12 weeks prior to screening
* pre-bronchodilator FEV1 60-85% at screening and other specified visits
* Post-bronchodilator reversibility >/=12%
* Non-smokers and prior smokers with no history of smoking within the past 12 months prior to screening and a total smoking history of ≤10 pack-years
* Subjects able to discontinue asthma medications for the duration of the study and be maintained using albuterol as required
* Body mass index between 18-40 kg/m2 inclusive

Key exclusion criteria include:

* Presence or recent history of any other active, severe, progressive, and/or uncontrolled clinical disease, eg, poorly controlled Type 1 or 2 diabetes, seizure disorder or epilepsy, cerebrovascular accident, significant cardiac conduction abnormalities
* Respiratory conditions other than asthma and allergic rhinitis, including but not limited to: severe nasal polyposis or chronic rhinosinusitis, chronic obstructive pulmonary disease, bronchiectasis, Churg-Strauss Disease, lung resection, pulmonary fibrosis (primary or secondary), pulmonary hypertension, cystic fibrosis, sarcoidosis
* History of life-threatening asthma, defined as a history of asthma episode(s) requiring intubation, and/or associated with hypercapnia; respiratory arrest or hypoxic seizures, asthma related syncopal episode(s)
* In patient hospitalization (not including ER visits) for an asthma exacerbation within the past year or during the run in period
* An asthma exacerbation requiring change in asthma therapy or oral/IV corticosteroids in the 3 months prior to screening
* History of seasonally unstable asthma where the season will coincide with the subject's participation in the study
* Use of prescription or non-prescription drugs, including beta blockers, tricyclic antidepressants, oral decongestants, benzodiazepines, digitalis, phenothiazines, monoamine oxidase inhibitors, etc
* Suspected hypersensitivity to the study drugs (including lactose) or severe milk protein allergy
* Clinically significant abnormalities in the screening ECG
* Evidence of alcohol or drug abuse or dependency within 6 months prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1128 (Actual)
Dates: Start 2014-10; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dik WH Ng, PhD, Study Director — Mylan Pharma UK Ltd.
Locations (101):
- United States (101):
  - Mylan Investigative Site #1, Birmingham, Alabama
  - Mylan Investigative Site #2, Little Rock, Arkansas
  - Mylan Investigative Site #3, Anaheim, California
  - Mylan Investigative Site #4, Bakersfield, California
  - Mylan Investigative Site #5, Burbank, California
  - Mylan Investigative Site #6, Costa Mesa, California
  - Mylan Investigative Site #7, Encinitas, California
  - Mylan Investigative Site #8, Fresno, California
  - Mylan Investigative Site #9, Fullerton, California
  - Mylan Investigative Site #10, Huntington Beach, California
  - Mylan Investigative Site #11, Huntington Beach, California
  - Mylan Investigative Site #12, Los Angeles, California
  - Mylan Investigative Site #13, Los Angeles, California
  - Mylan Investigative Site #14, Los Angeles, California
  - Mylan Investigative Site #15, Mission Viejo, California
  - Mylan Investigative Site #16, Napa, California
  - Mylan Investigative Site #17, Orange, California
  - Mylan Investigative Site #18, Riverside, California
  - Mylan Investigational Site #27, Rolling Hills Estates, California
  - Mylan Investigative Site #19, Sacramento, California
  - Mylan Investigative Site #20, San Diego, California
  - Mylan Investigative Site #21, San Jose, California
  - Mylan Investigative Site #101, Centennial, Colorado
  - Mylan Investigative Site #22, Centennial, Colorado
  - Mylan Investigative Site #23, Colorado Springs, Colorado
  - Mylan Investigative Site #24, Colorado Springs, Colorado
  - Mylan Investigative Site #25, Denver, Colorado
  - Mylan Investigative Site #26, Wheat Ridge, Colorado
  - Mylan Investigative Site #28, Coral Gables, Florida
  - Mylan Investigative Site #29, Gainesville, Florida
  - Mylan Investigative Site #30, Hialeah, Florida
  - Mylan Investigative Site #31, Largo, Florida
  - Mylan Investigative Site #32, Miami, Florida
  - Mylan Investigative Site #34, Miami, Florida
  - Mylan Investigative Site #33, Miami, Florida
  - Mylan Investigative Site #35, Miami, Florida
  - Mylan Investigative Site #36, New Port Richey, Florida
  - Mylan Investigative Site #37, Tallahassee, Florida
  - Mylan Investigative Site #38, Lawrenceville, Georgia
  - Mylan Investigative Site #39, River Forest, Illinois
  - Mylan Investigative Site #40, Shiloh, Illinois
  - Mylan Investigative Site #41, Lenexa, Kansas
  - Mylan Investigative Site #42, Bangor, Maine
  - Mylan Investigative Site #43, Baltimore, Maryland
  - Mylan Investigative Site #44, Bethesda, Maryland
  - Mylan Investigative Site #45, Wheaton, Maryland
  - Mylan Investigative Site #46, White Marsh, Maryland
  - Mylan Investigative Site #47, Fall River, Massachusetts
  - Mylan Investigative Site #48, North Dartmouth, Massachusetts
  - Mylan Investigative Site #49, North Dartmouth, Massachusetts
  - Mylan Investigative Site #50, Minneapolis, Minnesota
  - Mylan Investigative Site #51, Columbia, Missouri
  - Mylan Investigative Site #52, Rolla, Missouri
  - Mylan Investigative Site #53, St Louis, Missouri
  - Mylan Investigative Site #54, Warrensburg, Missouri
  - Mylan Investigative Site #55, Bozeman, Montana
  - Mylan Investigative Site #56, Missoula, Montana
  - Mylan Investigative Site #57, Bellevue, Nebraska
  - Mylan Investigative Site #58, Brick, New Jersey
  - Mylan Investigative Site #59, Ocean City, New Jersey
  - Mylan Investigative Site #60, Skillman, New Jersey
  - Mylan Investigative Site #61, New York, New York
  - Mylan Investigative Site #62, Asheville, North Carolina
  - Mylan Investigative Site #63, Charlotte, North Carolina
  - Mylan Investigative Site #64, Raleigh, North Carolina
  - Mylan Investigative Site #65, Canton, Ohio
  - Mylan Investigative Site #66, Cincinnati, Ohio
  - Mylan Investigative Site #67, Cincinnati, Ohio
  - Mylan Investigative Site #68, Sylvania, Ohio
  - Mylan Investigative Site #69, Toledo, Ohio
  - Mylan Investigative Site #70, Oklahoma City, Oklahoma
  - Mylan Investigative Site #71, Tulsa, Oklahoma
  - Mylan Investigative Site #72, Eugene, Oregon
  - Mylan Investigative Site #73, Lake Oswego, Oregon
  - Mylan Investigative Site #74, Medford, Oregon
  - Mylan Investigative Site #75, Portland, Oregon
  - Mylan Investigative Site #76, Jenkintown, Pennsylvania
  - Mylan Investigative Site #77, Pittsburgh, Pennsylvania
  - Mylan Investigative Site #78, Smithfield, Pennsylvania
  - Mylan Investigative Site #79, Providence, Rhode Island
  - Mylan Investigative Site #80, Warwick, Rhode Island
  - Mylan Investigative Site #81, North Charleston, South Carolina
  - Mylan Investigative Site #82, Spartanburg, South Carolina
  - Mylan Investigative Site #83, Spartanburg, South Carolina
  - Mylan Investigative Site #84, Boerne, Texas
  - Mylan Investigative Site #85, Dallas, Texas
  - Mylan Investigative Site #86, Dallas, Texas
  - Mylan Investigative Site #87, Dickinson, Texas
  - Mylan Investigative Site #88, El Paso, Texas
  - Mylan Investigative Site #89, New Braunfels, Texas
  - Mylan Investigative Site #90, San Antonio, Texas
  - Mylan Investigative Site #91, San Antonio, Texas
  - Mylan Investigative Site #92, Waco, Texas
  - Mylan Investigative Site #93, Provo, Utah
  - Mylan Investigative Site #94, South Burlington, Vermont
  - Mylan Investigative Site #95, Henrico, Virginia
  - Mylan Investigative Site #96, Seattle, Washington
  - Mylan Investigative Site #97, Spokane, Washington
  - Mylan Investigative Site #98, Tacoma, Washington
  - Mylan Investigative Site #99, Tacoma, Washington
  - Mylan Investigative Site #100, Greenfield, Wisconsin

REFERENCES:
- [Result] Ng D, Kerwin EM, White MV, Miller SD, Haughie S, Ward JK, Allan R. Clinical Bioequivalence of Wixela Inhub and Advair Diskus in Adults With Asthma. J Aerosol Med Pulm Drug Deliv. 2020 Apr;33(2):99-107. doi: 10.1089/jamp.2019.1547. Epub 2019 Oct 31. PMID 31634023

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MGR001 | Advair Diskus | Placebo
Started | 512 | 513 | 103
Completed | 499 | 500 | 98
Not Completed | 13 | 13 | 5
Not completed — Adverse Event | 4 | 4 | 4
Not completed — Lost to Follow-up | 3 | 5 | 1
Not completed — Withdrawal by Subject | 6 | 3 | 0
Not completed — Randomized in error (not treated) | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The baseline analysis population included all subjects who were randomized and received at least one dose of double-blind study medication. One subject was randomized in error to the Advair Diskus group but was not treated and so not included in the baseline analysis population
Groups:
- Total: Total of all reporting groups
Arm/Group | MGR001 | Advair Diskus | Placebo | Total
Number analyzed (Participants) | 512 | 512 | 103 | 1127
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.6 (14.08) | 42.5 (14.21) | 43.5 (13.85) | 42.6 (14.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 306 | 309 | 64 | 679
  Male | 206 | 203 | 39 | 448
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 102 | 92 | 24 | 218
  Not Hispanic or Latino | 410 | 420 | 79 | 909
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 11 | 11 | 1 | 23
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1 | 2
  Black or African American | 92 | 98 | 22 | 212
  White | 378 | 372 | 73 | 823
  More than one race | 30 | 31 | 6 | 67
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 512 | 512 | 103 | 1127
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 29.38 (6.026) | 29.12 (5.886) | 29.37 (5.890) | 29.26 (5.947)

OUTCOME MEASURES:

1. Primary Outcome: Forced Exhaled Volume in 1 Sec (FEV1) Area Under the Effect Curve on Day 1 (Assay Sensitivity)
Description: The FEV1 AUEC(0-12) on Day 1 was calculated from FEV1 measurements collected 30 minutes prior to morning dose, 0 minutes prior to morning dose, and at 0.5, 1, 2, 3, 4, 6, 8, 10, and 12 hours following completion of dosing on Day 1 (Visit 3). The baseline for the FEV1 AUEC(0-12) endpoint was the mean of the 2 predose FEV1 measures. To confirm assay sensitivity, both active treatments (MGR001 and Advair Diskus) had to be significantly superior to placebo
Time Frame: 0-12 hours after dosing on Day 1
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: L*hr
Arm/Group | MGR001 | Advair Diskus | Placebo
Number analyzed (Participants) | 508 | 510 | 102
L*hr | 3.9534 (0.1609) | 3.4964 (0.1595) | 0.8191 (0.3477)
Statistical Analysis 1: Comparison: MGR001 vs Placebo; MGR001 (Test) vs Placebo; Test type: Superiority — In order for the bioequivalence results to be valid, assay sensitivity had to be established. For assay sensitivity, the following comparisons were performed using the Full Analysis Set for each co-primary endpoint: MGR001 versus placebo, and Advair Diskus versus placebo. Assay sensitivity was demonstrated if the p-values for active treatment versus placebo were less than 0.05; p < 0.0001, ANCOVA
Statistical Analysis 2: Comparison: Advair Diskus vs Placebo; Advair Diskus (Reference) vs Placebo; Test type: Superiority — In order for the bioequivalence results to be valid, assay sensitivity had to be established.For assay sensitivity, the following comparisons were performed using the Full Analysis Set for each co-primary endpoint: MGR001 versus placebo, and Advair Diskus versus placebo. Assay sensitivity was demonstrated if the p-values for active treatment versus placebo were less than 0.05; p < 0.0001, ANCOVA

2. Primary Outcome: Forced Exhaled Volume in 1 Sec (FEV1) Area Under the Effect Curve on Day 1 (Bioequivalence)
Description: The FEV1 AUEC(0-12) on Day 1 was calculated from FEV1 measurements collected 30 minutes prior to morning dose, 0 minutes prior to morning dose, and at 0.5, 1, 2, 3, 4, 6, 8, 10, and 12 hours following completion of dosing on Day 1 (Visit 3). The baseline for the FEV1 AUEC(0-12) endpoint was the mean of the 2 predose FEV1 measures
Time Frame: 0-12 hours after dosing on Day 1
Population: Per Protocol Set
Measure: Least Squares Mean (Standard Error); unit: L*hr
Arm/Group | MGR001 | Advair Diskus | Placebo
Number analyzed (Participants) | 497 | 494 | 94
L*hr | 3.9734 (0.1704) | 3.5411 (0.1593) | 0.8400 (0.2983)
Statistical Analysis 1: Comparison: MGR001 vs Advair Diskus; Equivalence of MGR001 and Advair Diskus is established if the ratio of the LS means and 90% confidence interval are wholly contained within the interval 0.80-1.25 (i.e., 80%-125%); Test type: Equivalence — A linear analysis of covariance (ANCOVA) model was fitted for the endpoint and least-squares (LS) means were derived for each treatment. To assess equivalence, LS means (one for Test and one for Reference) from the ANCOVA models were used to generate Test/Reference ratios and 90% CIs were calculated by using Fieller's theorem. To demonstrate equivalence, the 90% CIs were each required to be wholly contained within the interval 0.80-1.25 (i.e., 80%-125%); Ratio (MGR001/Advair Diskus) = 1.120, 90% CI 2-sided [1.016 to 1.237] — Bioequivalence was established between active treatments (MGR001 and Advair Diskus) for the FEV1 AUEC0-12 clinical endpoint

3. Primary Outcome: FEV1 Trough Value (Assay Sensitivity)
Description: Change from baseline in trough (pre-dose) FEV1 at Day 29 was based on 2 pre-dose FEV1 assessments performed 30 minutes apart on Day 29. Baseline was calculated by taking the mean of [prebronchodilator FEV1 measured at a run-in visit and the mean of 2 predose FEV1 measures taken at Day 1]. To confirm assay sensitivity, both active treatments (MGR001 and Advair Diskus) had to be significantly superior to placebo.
Time Frame: Day 1 and Day 29
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: L
Arm/Group | MGR001 | Advair Diskus | Placebo
Number analyzed (Participants) | 504 | 505 | 100
L | 0.2927 (0.0162) | 0.2720 (0.0161) | 0.0575 (0.0353)
Statistical Analysis 1: Comparison: MGR001 vs Placebo; MGR001 (Test) vs Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.0001, ANCOVA
Statistical Analysis 2: Comparison: Advair Diskus vs Placebo; Advair Diskus (Reference) vs Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.0001, ANCOVA

4. Primary Outcome: FEV1 Trough Value (Bioequivalence)
Description: Change from baseline in trough (pre-dose) FEV1 at Day 29 was based on 2 pre-dose FEV1 assessments performed 30 minutes apart on Day 29. Baseline was calculated by taking the mean of [prebronchodilator FEV1 measured at a run-in visit and the mean of 2 predose FEV1 measures taken at Day 1]
Time Frame: Day 1 and Day 29
Population: Per Protocol Set
Measure: Least Squares Mean (Standard Error); unit: L
Arm/Group | MGR001 | Advair Diskus | Placebo
Number analyzed (Participants) | 498 | 497 | 99
L | 0.2911 (0.0163) | 0.2728 (0.0162) | 0.0574 (0.0355)
Statistical Analysis 1: Comparison: MGR001 vs Advair Diskus; [analysis description as in outcome 2, analysis 1]; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; Ratio (MGR001/Advair Diskus) = 1.069, 90% CI 2-sided [0.938 to 1.220] — Bioequivalence was established between active treatments (MGR001 and Advair Diskus) for change from baseline in trough FEV1 endpoint on Day 29

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from the signing of the ICF but are reported from Day 1 to 30 days after the last dose of double-blind study medication.
Description: Subjects were routinely queried for AEs using open-ended questions. Spontaneously reported AEs were also recorded. The most frequent AEs occurring in at least 3 subjects across the 3 treatment groups are reported, equating to 0.2% of subjects in the Safety Set.
Arm/Group | MGR001 | Advair Diskus | Placebo
All-Cause Mortality (participants affected / at risk) | 0/512 | 0/512 | 0/103
Serious Adverse Events (participants affected / at risk) | 0/512 | 0/512 | 0/103
Other Adverse Events (participants affected / at risk) | 39/512 | 51/512 | 10/103
OTHER ADVERSE EVENTS (reported when occurring in more than 0.2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MGR001 (N=512) | Advair Diskus (N=512) | Placebo (N=103)
Upper respiratory tract infection (Infections and infestations) | 7 | 11 | 0
Nasopharyngitis (Infections and infestations) | 3 | 7 | 2
Sinusitis (Infections and infestations) | 3 | 3 | 1
Oral candidiasis (Infections and infestations) | 4 | 2 | 0
Urinary tract infection (Infections and infestations) | 2 | 2 | 0
Viral upper respiratory tract (Infections and infestations) | 1 | 3 | 0
Bronchitis (Infections and infestations) | 2 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 3 | 0
Viral infection (Infections and infestations) | 1 | 2 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 7 | 10 | 5
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 5 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 2 | 0
Headache (Nervous system disorders) | 3 | 5 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes